CLINICAL TRIAL: NCT00187031
Title: A Phase II Study of Topotecan in Children With Recurrent Wilms Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: GlaxoSmithKline (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Monika Metzger, MD, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WILTOP
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Wilms Tumor
Keywords: Wilms Tumor
MeSH Terms: conditions — Wilms Tumor | interventions — Topotecan; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Topotecan, Filgrastim (G-CSF), Pegfilgrastim

INTERVENTIONS:
Drug: Topotecan, Filgrastim (G-CSF), Pegfilgrastim — See detailed description section for additional details.

SUMMARY:
In spite of the overall success of treating Wilms tumor, certain patients still have poor clinical outcomes. The sub-optimal outcomes for patients with anaplastic histology and recurrent Wilms tumor warrant the identification of new therapeutic agents. The objective of this trial is to estimate the response rate to two cycles of intravenous topotecan in children with recurrent Wilms tumor of favorable histology that is refractory to standard curative therapy.

DETAILED DESCRIPTION:
Topotecan administered intravenously over 30 minutes daily for 5 consecutive days for 2 consecutive weeks, with a two-day rest given in between the five-day treatment blocks. The topotecan dose started at 1.8 mg/m2/dosage and adjusted to attain a target systemic exposure of 80 plus or minus 10 ng-hr/ml.each cycle consists of 28 days and subsequent cycles can be administered upon hematological recovery. Patients with a CR, PR, or SD, can continue to receive up to a total of six cycles. Patients with PD are removed from the study.

Secondary Objectives include:

* To describe the anti-tumor activity of topotecan in children with recurrent Wilms tumor of anaplastic histology.
* To assess the relation between CYP3A4/5 genotype and the pharmacokinetics and pharmacodynamics of topotecan.
* To assess the relation between ABCG2 genotype and the pharmacokinetics and pharmacodynamics of topotecan.

ELIGIBILITY:
Inclusion Criteria:

* Favorable histology Wilms tumor that has recurred or progressed after primary treatment and at least one standard salvage treatment regimen OR anaplastic histology Wilms tumor that has recurred or progressed after primary treatment
* Age< 21 years of age at the time of study entry
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Adequate performance status

Exclusion Criteria:

* Subject is pregnant
* Subject is lactating
* Renal tumors other than Wilms tumors

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2002-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial response as per RECIST criteria). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Monika Metzger, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (7):
- United States (4):
  - Children's Healthcare, Atlanta, Georgia
  - Dana Farber, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Canada (3):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
  - Hospital of Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Metzger ML, Stewart CF, Freeman BB 3rd, Billups CA, Hoffer FA, Wu J, Coppes MJ, Grant R, Chintagumpala M, Mullen EA, Alvarado C, Daw NC, Dome JS. Topotecan is active against Wilms' tumor: results of a multi-institutional phase II study. J Clin Oncol. 2007 Jul 20;25(21):3130-6. doi: 10.1200/JCO.2007.10.9298. PMID 17634492
- See also: St. Jude Children's Research Hospital — http://www.stjude.org